CLINICAL TRIAL: NCT00634062
Title: Study of Lamotrigine Treatment of Affective Instability in Borderline Personality Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: D. Bradford Reich, M.D., McLean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-P-002640
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Borderline Personality Disorder
Keywords: Affective Lability; Borderline Personality Disorder; Pharmacotherapy
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Lamotrigine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — Subject in active active drug group will receive lamotrigine tablets 12.5 per day for the first week of the study. Dose of lamotrigine can be increased to 25mg per day during the second week of the study and may be increased each week thereafter for the next 9 weeks by 25mg per day. Subjects in active treatment group will receive lamotrigine for total of 12 weeks
  Other Names: Lamictal
  Arms: 1
Drug: Placebo — Subjects will receive 12.5mg of inert placebo per day during the first week of the study. Inert placebo can be increased to 25mg per day during the second week of the study and by 25mg per day each week for the next 9 weeks. Subjects can receive a total of 12 weeks of placebo.
  Arms: 2

SUMMARY:
This study investigates the hypothesis that instability in mood in patients with borderline personality disorder will respond the mood stabilizing medication lamotrigine.

DETAILED DESCRIPTION:
Affective instability is one of the most prominent symptoms in borderline personality disorder. Currently there are no prospective studies of treatment of this symptom with mood stabilizing medications. This study examines the effectiveness of lamotrigine compared to placebo in reducing emotional instability of several types in borderline patients. The types of emotional instability studied involve anger, anxiety, depression, and elation. Subjects entering this 12 week study will be blind to whether they are receiving active medication or placebo. They will be asked to report levels of instability in their mood on a weekly basis. They will also be asked weekly to rate the intensity of other symptoms of borderline personality disorder symptoms, such as unstable relationships, self-harm, and impulsive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Borderline Personality Disorder with high levels of emotional instability

Exclusion Criteria:

* Clinical diagnosis of Bipolar Disorder
* Clinical diagnosis of psychiatric disorder related to general medical condition
* Clinical diagnosis of substance abuse disorder within the last 60 days
* Clinical diagnosis of psychotic disorder
* Previous treatment with lamotrigine
* Pregnancy or nursing
* Currently hospitalized
* Active suicidal or homicidal ideation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Changes in score of Affective Lability Scale | Baseline and then weekly for 12 weeks
Changes in the score of the Affective Lability Item of the Zanarini Rating Scale for Borderline Personality Disorder | Baseline and then weekly for 12 weeks

SECONDARY OUTCOMES:
Scores of individual items on the Zanarini Rating Scale for Borderline Personality Disorder | Baseline and then weekly for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: D. Bradford Reich, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Weinstein W, Jamison KL. Retrospective case review of lamotrigine use for affective instability of borderline personality disorder. CNS Spectr. 2007 Mar;12(3):207-10. doi: 10.1017/s1092852900020927. PMID 17329981
- [Background] Tritt K, Nickel C, Lahmann C, Leiberich PK, Rother WK, Loew TH, Nickel MK. Lamotrigine treatment of aggression in female borderline-patients: a randomized, double-blind, placebo-controlled study. J Psychopharmacol. 2005 May;19(3):287-91. doi: 10.1177/0269881105051540. PMID 15888514
- [Background] Pinto OC, Akiskal HS. Lamotrigine as a promising approach to borderline personality: an open case series without concurrent DSM-IV major mood disorder. J Affect Disord. 1998 Dec;51(3):333-43. doi: 10.1016/s0165-0327(99)00007-5. PMID 10333987
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174